CLINICAL TRIAL: NCT00155441
Title: Effects of Cognitive-Behavioral Therapy on Sleep Disturbance in Peritoneal Dialysis Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Far Eastern Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9461700509
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2005-05

CONDITIONS: Sleep Disorders; Kidney Diseases
Keywords: sleep disorder; peritoneal dialysis; cognitive-behavioral therapy; sleep disorder:C23.888.592.796; peritoneal dialysis: F03.870.664
MeSH Terms: conditions — Sleep Wake Disorders; Kidney Diseases | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: cognitive-behavioral therapy

SUMMARY:
Sleep disturbance is prevalent in chronic dialysis patients and there is a negative correlation between the quality of life and overall survival and sleep disturbance in them. Cognitive-behavioral therapy is an effective behavioral therapy for insomnia clinically. In previous studies, cognitive-behavioral therapy can redress anxiety in chronic hemodialysis patients. This study tries to elucidate its therapeutic effect on the sleep disturbance in chronic peritoneal dialysis patients.

DETAILED DESCRIPTION:
Sleep disturbance is prevalent in chronic dialysis patients and there is a negative correlation between the quality of life and overall survival and sleep disturbance in them. So many factors interfering the sleep of these patients, however, there is no effective therapy for them except some drugs, such as hypnotics or anxiolytics. Cognitive-behavioral therapy is an effective behavioral therapy for insomnia clinically and it contains three therapeutic domains including stimulus control, sleep restriction therapy, and relaxation training. It has been proven to be beneficial in improving sleep pattern in chronic insomnia and cancer patients and alcoholism. In previous studies, cognitive-behavioral therapy can redress anxiety in chronic hemodialysis patients, however, there is no clinical evidence revealing its effectiveness upon sleep disorders in hemodialysis and peritoneal dialysis patients. Our study tries to elucidate the therapeutic effect of cognitive-behavioral therapy on the sleep disturbance in chronic peritoneal dialysis patients.

We will perform cognitive-behavioral therapy to eligible peritoneal dialysis patients and evaluate the sleep condition before and after the therapy. Moreover, clinical conditions, biochemical and hematological parameters, inflammatory mediators in blood will be measured at baseline, before and after therapy.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing peritoneal dialysis (PD) for at least 3 months
* Older than 18 years
* Have sleep disturbance subjectively

Exclusion Criteria:

* Unstable clinical conditions or evidence of malignancy
* Pregnancy
* Participation in another study that would interfere with the outcome of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-06

PRIMARY OUTCOMES:
Check Pittsburgh Sleep Quality Index and restless leg syndrome index: in 1st and 3rd months

SECONDARY OUTCOMES:
The hematologic, biochemical markers, and peritoneal function in 1st and 3rd months

CONTACTS AND LOCATIONS:
Overall Officials: Tun-Jun Tsai, Ph.D., M.D., Principal Investigator — Division of Nephrology, Department of Internal Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Dawan, Taiwan

REFERENCES:
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553